CLINICAL TRIAL: NCT03952780
Title: Korean Registry of Percutaneous EVAR With INCRAFT Stent Graft for the Treatment of Abdominalaortic Aneurysm (K-INCRAFT)
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2018-0081
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: abdominal aortic aneurysm; endovascular repair; stent graft
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The sudy purpose is to investigate efficacy and safety of percutaneous endovascular aortic aneurysm repair using INCRAFT stent graft for Korean patients with abdominal aortic aneurysm. This study is designed as an investigator-initiated, multi-center, single-arm, prospective registry study. A total of 100 patients who meet all inclusion criteria, but none of exclusion criteria will be enrolled after the implantation of INCRAFT stent graft. The primary efficacy outcome is technical success defined as successful deployment of the stent-graft with no type I/III endoleak, unintentional coverage of visceral aortic branches or internal iliac arteries at the end of the procedure, and with successful removal of the delivery system. The primary safety outcome is major vascular complications at 30 days including. The study subjects will be followed for 12 months.

DETAILED DESCRIPTION:
Prospective single-arm multicenter registry

ELIGIBILITY:
Inclusion Criteria:

* 1. AAA with one of following indications

  1. AAA with maximum diameter > 5 cm,
  2. AAA with maximum diameter > 4 cm with an increase >0.5 cm during the preceding 6 months
  3. Saccular type AAA irrespective of the sac diameter.
* 2. Proximal aortic neck length ≥10 mm with a diameter ≥ 17 and ≤ 31 mm in combination with supra- and infrarenal angulation ≤ 60 degree.
* 3. Iliac landing zone with a length ≥15 mm and a diameter ≥ 7 and ≤ 22 mm
* 4. Femoral access vessels should be adequate to fit the selected delivery system
* 5. Minimum overall AAA treatment length (proximal landing location to distal landing location to distal landing location) ≥128 mm
* 6. Aortic bifurcation >18 mm in diameter
* 7. Patents with age of 19-80 years.
* 8. Male or non-pregnant female
* 9. Voluntary participation in the study with signed informed consent form.

Exclusion Criteria:

* 1. Dissecting or ruptured abdominal aortic aneurysm
* 2. Presence of connective tissue disease (Marfan's syndrome or Ehlers-Danlos syndrome).
* 3. Prior AAA or iliac artery repair
* 4. Active infection or active vasculitis.
* 5. Myocardial infarction or cerebrovascular accident within 3 months prior to study enrolment.
* 6. Need for renal artery coverage (e.g. Chimney graft)
* 7. Dialysis-dependent renal failure or serum creatinine >2.0 mg/dl
* 8. Intolerance/hypersensitivity to contrast media or antiplatelet drugs.
* 9. Positive pregnancy test.
* 10. Participation in another medical research study within 1 month of study enrolment.
* 11. Planned concomitant surgical procedures (other than left subclavian artery transposition or bypass) or major surgery within 30 days of study enrolment.
* 12. Patients with life expectancy less than 1 year

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with abdominal aortic aneurysm treated with INCRAFT stent graft
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Technical success | At the end of the procedure
  Technical success defined as successful deployment of the stent-graft with no type I/III endoleak, unintentional coverage of visceral aortic branches or internal iliac arteries at the end of the procedure, and with successful removal of the delivery system. Primary conversion or additional implantation of bare metal stent, aortic cuff or EndoAnchors to treat type I endoleak is considered a technical failure.

SECONDARY OUTCOMES:
Major adverse event | 30 days
  Major adverse event, a composite of death, myocardial infarction, stroke, or renal failure requiring dialysis) at 30 days
Major adverse event | 1 year
  Major adverse event, a composite of death, myocardial infarction, stroke, or renal failure requiring dialysis) at 1 year
Aneurysm-related death | 30 days
  All-cause death at 30 days
Aneurysm-related death | 1 year
  All-cause death at 1 year
Aneurysm-related death | 30 days
  Aneurysm-related death at 30 days
Aneurysm-related death | 1 year
  Aneurysm-related death at 1 year
Reintervention | 1 year
  Reintervention at 1 year
Type I/III endoleaks | 30 days
  Type I/III endoleaks at 30 days
Type I/III endoleaks | 1 year
  Type I/III endoleaks at 1 year
Aneurysm-related event | 1 year
  Aneurysm-related event (aneurysm-related death, reintervention, and aorta expansion> 5 mm, device migration, conversion to open repair, stent graft fracture, stent graft occlusion) at 1 year
All vascular complications related to the INCRAFT device or aneurysm requiring surgical or endovascular interventions | 30 days
  All vascular complications at 30 days related to the INCRAFT device or aneurysm requiring surgical or endovascular interventions
Number of closure devices used for the closure of access sites. | 30 days
  Number of closure devices used for the closure of access sites.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University Health System, 50 Yonsei-ro, Seodaemun-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No